CLINICAL TRIAL: NCT03208283
Title: Evaluation of the Impact of Water Metsertion Phase of Flexible Sigmoidoscopy in the Training of Primary Care Doctors or Nurse Endoscopists for Colorectal Cancer Screening: A Randomized Controlled Study (FSW Study)
Brief Title: Evaluation of the Impact of Water Method During Insertion Phase of Flexible Sigmoidoscopy in Training
Acronym: FSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Associate Director of S.H. Ho Centre for Digestive Health, Institute of Digestive Disease, the Chinese University of Hong Kong, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FSW
Record Dates: First submitted 2017-05-15; First posted 2017-07-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer Screening
MeSH Terms: interventions — Pneumoradiography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Air insufflation group (Active Comparator): During the insertion phase of the initial 30 FS procedures, air insufflation will be used to allow passage of endoscope to ≥ 50cm above anal verge (including rectum, sigmoid colon and part of descending colon), or to the limit of patient tolerance of an unsedated procedure. Trainees will be allowed 10 minutes for the insertion phase. The unassisted portion of the examination would be terminated if reasonable progress is not being attained, excessive patient discomfort observed, or the supervising endoscopist believes that patient safety may be compromised. During the withdrawal phase, air insufflation will be used in standard fashion for examination of the colonic mucosa.
  Interventions: Diagnostic Test: Air insufflation group
- Water method group (Active Comparator): During the insertion phase of the initial 30 FS procedures, sterile water will be infused by a standard endoscopy water pump into the distal colon to allow passage of endoscope to ≥ 50cm above anal verge (including rectum, sigmoid colon and part of descending colon), or to the limit of patient tolerance of an unsedated procedure. Air insufflation will not be used during the insertion phase. Trainees will be allowed 10 minutes for the insertion phase. The unassisted portion of the examination would be terminated if reasonable progress is not being attained, excessive patient discomfort observed, or the supervising endoscopist believes that patient safety may be compromised. During the withdrawal phase, air insufflation will be used in standard fashion for examination of the colonic mucosa.
  Interventions: Diagnostic Test: Water method group

INTERVENTIONS:
Diagnostic Test: Water method group — During the insertion phase of the initial 30 FS procedures, sterile water will be infused by a standard endoscopy water pump into the distal colon to allow passage of endoscope to ≥ 50cm above anal verge (including rectum, sigmoid colon and part of descending colon), or to the limit of patient tolerance of an unsedated procedure. Air insufflation will not be used during the insertion phase. Trainees will be allowed 10 minutes for the insertion phase. The unassisted portion of the examination would be terminated if reasonable progress is not being attained, excessive patient discomfort observed, or the supervising endoscopist believes that patient safety may be compromised. During the withdrawal phase, air insufflation will be used in standard fashion for examination of the colonic mucosa.
  Other Names: Water Immersion
  Arms: Water method group
Diagnostic Test: Air insufflation group — During the insertion phase of the initial 30 FS procedures, air insufflation will be used to allow passage of endoscope to at least 50cm above anal verge (including rectum, sigmoid colon and part of descending colon), or to the limit of patient tolerance of an unsedated procedure. Trainees will be allowed 10 minutes for the insertion phase. The unassisted portion of the examination would be terminated if reasonable progress is not being attained, excessive patient discomfort observed, or the supervising endoscopist believes that patient safety may be compromised. During the withdrawal phase, air insufflation will be used in standard fashion for examination of the colonic mucosa.
  Other Names: Air insufflation
  Arms: Air insufflation group

SUMMARY:
Colonoscopy is a sedated procedure traditionally performed using air insufflation during the insertion phase of the procedure. Recently, the use of water method (eg, water infusion or water exchange techniques) during the insertion phase of colonoscopy has been reported to increase the proportion of patients in whom complete unsedated colonoscopy could be achieved, reduce patient recovery time burdens, decrease abdominal discomfort during and after colonoscopy, enhance cecal intubation, and increase willingness to repeat an unsedated colonoscopy. However, there has been no study on the use of water method during the training of primary care doctors or nurse endoscopists in flexible sigmoidoscopy for colorectal cancer screening.

In unsedated endoscopic procedure such as FS, endoscope insertion techniques that can potentially reduce patient discomfort and increase the rate of achieving an adequate depth of scope insertion are desirable. Our current study aims to evaluate the impact of water method during insertion phase of FS in the training of primary care doctors or nurse endoscopists for colorectal cancer screening.

DETAILED DESCRIPTION:
It is estimated that there are about 1.2 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence and mortality globally. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality.

CRC is one of the most preventable cancers because its development in general follows an adenoma-carcinoma sequence. Adenomas are considered precursor lesions for CRC. Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 50. Modalities such as guaiac-based fecal occult blood tests (gFOBT), fecal immunochemical tests (FIT), flexible sigmoidoscopy, and colonoscopy are among the acceptable options for CRC screening. Studies have shown that early detection and removal of colorectal adenoma by screening flexible sigmoidoscopy (FS) and screening colonoscopy with polypectomy reduce CRC incidence and mortality.

Approximately two-thirds of CRC are located in the sigmoid colon and rectum, which can be diagnosed by FS. In countries where colonoscopy may not be widely available or a prolonged waiting time exists, FS becomes an attractive option for CRC screening.

When compared to colonoscopy, FS has the advantages of being an unsedated procedure, requiring less stringent bowel prep, and being less technically demanding. While flexible sigmoidoscopy have traditionally been performed by gastroenterologists or surgeons, studies have demonstrated that adequately trained primary care doctors and nurse endoscopists can perform screening flexible sigmoidoscopy as safely and effectively as gastroenterologists or surgeons. The American Society for Gastrointestinal Endoscopy (ASGE), the Society of American Gastrointestinal Endoscopic Surgeons (SAGES), and the The Society of Gastrointestinal Nurses and Associates (SGNA) recommend 25 supervised procedures for training in FS. Hawes R et al reported that at least 30 supervised procedures were needed before 85% - 90% of the procedures were graded as competent in doctors without prior experience on rigid sigmoidoscopy. In another report, at least 50 supervised procedures have been suggested for FS training of clinicians without prior endoscopic skills.

From a technical standpoint, colonoscopy is a sedated procedure traditionally performed using air insufflation during the insertion phase of the procedure. Recently, the use of water method (eg, water infusion or water exchange techniques) during the insertion phase of colonoscopy has been reported to increase the proportion of patients in whom complete unsedated colonoscopy could be achieved, reduce patient recovery time burdens, decrease abdominal discomfort during and after colonoscopy, enhance cecal intubation, and increase willingness to repeat an unsedated colonoscopy. However, there has been no study on the use of water method during the training of primary care doctors or nurse endoscopists in flexible sigmoidoscopy for colorectal cancer screening.

In unsedated endoscopic procedure such as FS, endoscope insertion techniques that can potentially reduce patient discomfort and increase the rate of achieving an adequate depth of scope insertion are desirable. Our current study aims to evaluate the impact of water method during insertion phase of FS in the training of primary care doctors or nurse endoscopists for colorectal cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive asymptomatic patients suitable for CRC screening by FS
* Age 50 - 70 years
* Written informed consent available

Exclusion Criteria:

* Contraindications for endoscopy due to comorbidities
* Unable to provide written informed consent
* Personal history of polyposis syndrome, personal history of CRC, personal history of inflammatory bowel disease
* Coagulopathy (INR>1.5) or thrombocytopenia (platelets <50,000)
* Pregnant patients

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-10-28 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Independently performed flexible sigmoidoscopy completion rate by each trainee | 12 weeks
  The percentage of unassisted FS procedure completed within the allowed 10 minutes in the initial 30 FS procedures for each trainee endoscopist
The mean independently performed flexible sigmoidoscopy completion rate in each study group | 12 weeks
  2) The mean percentage of unassisted FS procedure completed within the allowed 10 minutes in the initial 30 FS procedures by all trainee endoscopists in the air insufflation group, and the water method group, respectively

SECONDARY OUTCOMES:
Polyp detection rate | 12 weeks
  Number and type of polyp detected during flexible sigmoidoscopy
Insertion distance | 12 weeks
  Mean unassisted scope insertion distance within the allowed 10 minutes and the total insertion distance in the initial 30 FS procedures
Procedural time | 12 weeks
  Mean insertion time, withdrawal time, and total procedure time in the initial 30 FS in each study group
Patients' satisfaction | 12 weeks
  This will be assessed by validated patient satisfaction questionnaire for gastrointestinal endoscopy (modified GHAA-9)

CONTACTS AND LOCATIONS:
Overall Officials: Shing Yan Raymond Tang, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Digestive Health, Institute of Digestive Disease, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No